CLINICAL TRIAL: NCT06306014
Title: Evaluation of EXL01, a New Live Biotherapeutic Product to Prevent Recurrence of Clostridioides Difficile Infection in High-risk Patients
Acronym: LIVEDIFF
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Exeliom Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL22_0980; 2023-506232-32-00 (Other: EU CT Number)
Record Dates: First submitted 2024-02-21; First posted 2024-03-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Clostridioides Difficile Infection; Recurrent Infection
Keywords: Clostridioides difficile Infection; Live Biotherapeutic Product; Microbiota; Recurrent Infection
MeSH Terms: conditions — Clostridium Infections; Reinfection

STUDY DESIGN:
Intervention Model Description: Part A = Single Arm open label. Part B = Randomised, placebo-controlled, double-blind.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A: None (Open-label). Part B: Double-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A (Open-Label EXL01) (Experimental)
  Interventions: Drug: EXL01
- Part B (EXL01) (Experimental)
  Interventions: Drug: EXL01
- Part B (Placebo) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EXL01 — Following a at least 10-days vancomycin treatment :
  Oral EXL01 including:
  * 10 capsules per day in week 1 and 2
  * 4 capsules per day, in weeks 3 and 4
  * 1 capsule per day in weeks 5 to 8 Phase I : EXL01 during a 8 weeks open-label period
  Arms: Part A (Open-Label EXL01)
Drug: EXL01 — Following a at least 10-days vancomycin treatment :
  Oral EXL01 including:
  * 10 capsules per day in week 1 and 2
  * 4 capsules per day, in weeks 3 and 4
  * 1 capsule per day in weeks 5 to 8 Phase II: EXL01 during a 8 weeks double blind placebo-controlled period
  Arms: Part B (EXL01)
Drug: Placebo — Following a at least 10-days vancomycin treatment:
  Oral placebo including:
  * 10 capsules per day in week 1 and 2
  * 4 capsules per day, in weeks 3 and 4
  * 1 capsule per day in weeks 5 to 8 Phase II : Placebo during a 8 weeks double blind placebo-controlled period
  Arms: Part B (Placebo)

SUMMARY:
Clostridioides difficile infection (CDI) is the leading cause of nosocomial diarrhea in Europe, with over 120,000 cases and almost 3,700 deaths per year. This infection is characterized by a high risk of recurrence after cure, ranging from almost 20% after a first episode to over 60% after 2 recurrences, or in the case of specific risk factors.

Currently, first-line treatment of CDI is based on oral antibiotics such as fidaxomicin or vancomycin. These antibiotic treatments, which are effective in 89% and 86% of first-episode cases respectively, do not correct the microbiological imbalance underlying the onset of CDI and may, on the contrary, encourage recurrence by contributing to the maintenance of a deleterious change in the microbiota (dysbiosis) through the elimination of bacteria other than C. difficile, due to their spectrum of activity. In a number of patients, this ecological imbalance can no longer be restored after antibiotic treatment, leading to multiple recurrences of CDI.

In this context, fecal microbiota transplantation (FMT) has been validated for over 10 years for the prevention of recurrence in multi-recurrent CDI. The principle of FMT is based on the use of a pharmaceutical preparation made from the stool of a healthy donor, administered within the digestive tract of a patient for therapeutic purposes.

Currently, in the case of multiple recurrences, it is the recommended first-line treatment (from 2 recurrences) and the most effective, with a clinical efficacy preventing recurrence of CDI in 69% to 89% of cases at 8 weeks post-treatment, with a good safety profile.

Among the microbial factors promoting CDI, the loss of the bacterial species Faecalibacterium prausnitzii constitutes a specific therapeutic target. F. prausnitzii is a commensal bacterium of the human gut, making up nearly 5% of the fecal microbiota, and has been shown to be associated with an individual's state of health. A drop in its relative abundance is associated with an increased risk of numerous diseases, such as Crohn's disease and colorectal cancer. In CDI, F prausnitzii is greatly diminished. Moreover, low abundance of F. prausnitzii is predictive of C. difficile recurrence. Its abundance in stools is increased after FMT and is also predictive of response to treatment. From a pathophysiological point of view, one of the preventive effects of F. prausnitzii on recurrence would be mediated by its ability to hydrolyze the bile acids involved in the germination of C. difficile spores.

The aim of this Phase I/II trial is to assess the efficacy and safety of oral administration of EXL01, a single isolated unmodified strain of F. prausnitzii, in preventing CDI recurrence in high-risk patients at W8. The study will be conducted in 2 parts. The phase I (Part A) is planned to include 6 patients. The phase II (Part B) will include 50 patients in two arms (25 patients respectively in the placebo and EXL01 arm).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥18 years of age
* ≥3rd episode of proven C. difficile infection (≥3 liquid stools per day and detection of toxigenic C. difficile in stool by PCR or enzyme-linked immunosorbent assay or immunochromatography or toxigenic culture) within 6 months with an interval ≤ 12 weeks since the end of treatment of the previous episode of resolved CDI or 2nd episode of proven C. difficile infection (≥3 liquid stools per day and detection of toxigenic C. difficile in the stools by PCR or enzyme-linked immunosorbent assay or immunochromatography or toxigenic culture) within 6 months with an interval ≤ 12 weeks since the end of treatment of the previous episode of resolved CDI with at least one of the following risk factors:

  * Age ≥70 years
  * Chronic renal failure (haemodialysis or GFR<60ml/min
  * History of severe or severe-complicated CDI (excluding current episode) according to ESCMID 2021 criteria
  * ≥3 CDI in the last 12 months (including current episode)
  * CDI associated with care defined as CDI occurring during hospitalisation (<3 months)
* On current or planned vancomycin treatment per os
* Patient able to give free, informed and written consent
* Enrolled in compulsory national social security scheme

Exclusion Criteria:

* Currently participating or has participated in a study with an investigational compound or device within 3 months prior to the first dose of the study intervention.
* Severe C. difficile infection severe (defined by the presence of a white blood cell count >15×10⁹ cells/L or a body temperature >38.5°C or >50% increase in the patient's baseline creatinine related to CDI at the time of V1) and/or complicated (defined by any of the factors attributed to current Clostridioides difficile infection (CDI): hypotension, septic shock, elevated serum lactate, ileus, toxic megacolon, intestinal perforation or any fulminant course of the disease)
* Refractory C. difficile infection defined as lack of response to well-conducted per os vancomycin or fidaxomicin treatment with ≥3 liquid stools per day after ≥5 days of treatment
* Cirrhosis with Child C score
* Hospitalization in continuing care unit or intensive care unit
* Immunosuppression including :

  * Malignant hemopathy under treatment (excluding CLL)
  * HIV AIDS stage
  * Stem cell allograft ≤ 12 months
  * Aplasia (<500 PNN/mm3) at inclusion
  * Treatment with >20mg prednisone equivalent within 14 days prior to inclusion (excluding inhaled or topical treatment).
* Personal history of gastrointestinal resection other than appendectomy (gastrectomy, esophagectomy, colonic or small bowel resection, short small bowel syndrome).
* Personal history of small intestinal microbial overgrowth
* Inflammatory bowel disease
* Proven celiac disease
* Current stoma (ileostomy or colostomy) or within the last 6 months, or any other intra-abdominal surgery within the 3 months prior to treatment
* major surgery or trauma ≤ 4 weeks before the start of treatment
* Antibiotic therapy in progress or planned during the study for an infection other than CDI
* Surgery scheduled during the study requiring perioperative antibiotics.
* -Women without contraception*, pregnant or breastfeeding women
* History of hypersensitivity to EXL01 and/or to any of its excipients (D-mannitol, sucrose, maltodextrin, L-cysteine, L-cysteine hydrochloride, magnesium stearate and hydroxypropylmethylcellulose), and/or to soy or soy-containing products.
* History of hypersensitivity to vancomycin as mentioned in local prescribing information.
* Personal history of fecal microbiota transplantation < 12 months
* Persons deprived of liberty by judicial or administrative decision
* Adults under legal protection or unable to give consent
* Swallowing disorders making oral treatment impossible
* Participation in another interventional study within 3 months prior to inclusion. (Patients who have entered the follow-up phase of an interventional study may participate provided that more than 3 months have elapsed since the last intervention).
* Expected life expectancy of less than 6 months
* Presents a known psychiatric disorder that would interfere with adequate cooperation with study requirements.
* Regular use of illicit or recreational drugs
* Anticipated administration during the study of treatment that is expected to cause diarrhea (chemotherapy, colonic preparation prior to colonoscopy)
* History of chronic diarrhea (> 3 watery stools per day for > 4 weeks) not related to gastrointestinal infection.
* Clinically significant medical or surgical condition not mentioned in the above criteria which, in the opinion of the investigator, could interfere with the administration of study drug, the interpretation of study safety or efficacy data, or compromise the safety or well-being of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-01-07 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | at Week 1, Week 2, Week 4, Week 8, Week 16
  Phase I The primary endpoint is the occurrence of serious adverse events (CTCAE grade≥3) during treatment and follow-up and discontinuation of treatment due to adverse events attributed to treatment
Evaluation of the efficacy of EXL01 in preventing recurrence of C. difficile infection in patients at high risk of recurrence | at Week 8
  Phase II The primary endpoint is the proportion of patients at W8 after the start of treatment who had a recurrence of toxigenic C. difficile defined by ≥3 liquid stools per day for more than 48 hours + detection of C. difficile toxin in stool (enzyme-linked immunosorbent assay or toxigenic culture +/- PCR) resulting in the initiation of CDI-specific treatment.

SECONDARY OUTCOMES:
Evaluation of the efficacy of EXL01 in preventing recurrence of C. difficile infection in patients at high risk of recurrence | at Week 8
  Phase I Proportion of patients at W8 after the start of treatment who had a recurrence of toxigenic C. difficile defined by ≥3 liquid stools per day for more than 48 hours + detection of C. difficile toxin in stool (enzyme-linked immunosorbent assay or toxigenic culture +/- PCR) resulting in the initiation of specific treatment for CDI.
Evaluation of the safety and tolerability profile of oral EXL01 | at Week 2, Week 4, Week 8, Week 16
  Phase II Occurrence of adverse events (CTCAE grade≥3) during treatment and follow-up, and discontinuation of treatment due to adverse events
Number of stools per day over the past 24 hours | at Week 0, Week 1, Week 2, Week 4, Week 8, Week 16
  Phase I Assessment of digestive symptoms during treatment and follow-up Digestive symptoms are measured at each visit using a stool calendar
Stool consistency, as assessed by the Bristol scale, over the past 24 hours | at Week 0, Week 1, Week 2, Week 4, Week 8, Week 16
  Phase I Digestive symptoms are measured at each visit using the stool calendar
Abdominal discomfort assessed by a validated irritable bowel syndrome scale | at Week 8, Week 16
  Phase I Assessment of digestive symptoms during treatment and follow-up Digestive symptoms are measured at each visit (IBS-SSS modified, GCSI, GERDQ)
Number of stools per day over the past 24 hours | at Week 0, Week 2, Week 4, Week 8, Week 16
  Phase II Assessment of digestive symptoms during treatment and follow-up Digestive symptoms are measured at each visit using a stool calendar
Stool consistency, as assessed by the Bristol scale, over the past 24 hours | at Week 0, Week 2, Week 4, Week 8, Week 16
  Phase II Digestive symptoms are measured at each visit using the stool calendar
Abdominal discomfort assessed by a validated irritable bowel syndrome scale | at Week 8, Week 16
  Phase II Assessment of digestive symptoms during treatment and follow-up Digestive symptoms are measured at each visit (IBS-SSS modified, GCSI, GERDQ)
Assessment of patient quality of life during treatment and follow-up | At Week 8 and Week 16
  Phases I and II Patient quality of life at W8 and M4 measured by a validated digestive disease quality of life questionnaire (GIQLI)
Assessment of recurrence of C. difficile infection | At Week 16
  Phases I and II percentage of patients with recurrence of C. difficile infection at M4
Evaluation of the presence of EXL01 in the fecal microbiota | At Week 8
  Phases I and II Level of F. prausnitzii (qPCR) in stool at W8 versus W0
Assessment of EXL01 persistence in the intestinal microbiota | At Week 0 and Week 16
  Phases I and II Level of F. prausnitzii (qPCR) in stool at M4 versus W0
16S rRNA sequencing or shotgun | at Week 0, Week 1, Week 2, Week 4, Week 8, Week 16
  Phase I Gut microbiota composition at each visit
16S rRNA sequencing or shotgun | at Week 0, Week 2, Week 4, Week 8, Week 16
  Phase II Gut microbiota composition at each visit
Assessment of the persistence of toxigenic C. difficile in the stool of patients in clinical remission during the study. | at Week 0, Week 1, Week 2, Week 4, Week 8, Week 16
  Phase I Percentage of patients at each visit with a positive stool PCR test for toxigenic C. difficile considered to be in clinical remission
Assessment of the persistence of toxigenic C. difficile in the stool of patients in clinical remission during the study. | at Week 0, Week 2, Week 4, Week 8, Week 16
  Phase II Percentage of patients at each visit with a positive stool PCR test for toxigenic C. difficile considered to be in clinical remission
Assessment of recurrences of C. difficile infection requiring hospitalization | At Week 8
  phases I and II percentage of patients with recurrence of C. difficile infection requiring hospitalization at W8
Assessment of recurrences of C. difficile infection requiring hospitalization | at Week 16
  phases I and II percentage of patients with recurrence of C. difficile infection requiring hospitalization at M4
Assessment of recurrences of C. difficile infection requiring surgery | at Week 8
  phases I and II phases I and II percentage of patients with a recurrence of C. difficile infection requiring surgery at W8
Assessment of recurrences of C. difficile infection requiring surgery | at Week 16
  phases I and II percentage of patients with recurrent C. difficile infection requiring surgery at M4

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BENECH, MD, Principal Investigator — Hospices Civils de Lyon
Locations (9):
- France (9):
  - CH Annecy Genevois Service de Maladies infectieuses, Annecy
  - Service d'hépato-gastroentérologie - CHU Estaing, Clermont-Ferrand
  - CHU Grenoble Service Maladies infectieuses et tropicales, Grenoble
  - Service d'Hépato-gastroentérologie Hôpital de la Croix Rousse, Lyon
  - APHM La Timone Service de Maladies infectieuses, Marseille
  - Service d'hépato-gastroentérologie - Hôpital Saint Antoine (APHP), Paris
  - Service d'infectiologie - Hôpital Nord / CHU Saint Etienne, Saint-Etienne
  - Service de médecine interne - Pôle des maladies de l'appareil digestif - CHU de Toulouse, Toulouse
  - Service de Maladies Infectieuses - CH de Valence, Valence